CLINICAL TRIAL: NCT06378216
Title: Myotonic Dystrophy Type 1 Congenital and Juvenile Form: From Diagnosis to Rehabilitation
Brief Title: Myotonic Dystrophy Type 1 Congenital and Juvenile Form: From Diagnosis to Rehabilitation [MDCJ-NeuBeRe]
Acronym: MDCJ-NeuBeRe
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: MEDEA 975
Record Dates: First submitted 2024-03-19; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Myotonic Dystrophy 1
Keywords: Myotonic dystrophy congenital form; Myotonic dystrophy infantile form; neuropsychological evaluation; behavioral evaluation; brain imaging study
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myotonic Dystrophy type 1: Myotonic Dystrophy type 1 -congenital form Myotonic Dystrophy type 1-infantile form
  Interventions: Diagnostic Test: neurocognitive evaluations

INTERVENTIONS:
Diagnostic Test: neurocognitive evaluations — clinical and neurocognitive evaluations neuroradiological evaluation through cerebral magnetic resonance
  Other Names: cerebral imaging

SUMMARY:
The rationale of the study is to collect structured data in the neuropsychological, clinical neuroradiologic and neurorehabilitation fields in children/young people affected by congenital and juvenile myotonic dystrophy. Children affected by the congenital form (CDM1) present important brain alterations present since birth while, on the contrary, patients with the adult form of DM1 often present a degenerative, slowly progressive neurocognitive picture. Promising therapies that aim to correct the molecular mechanism underlying the symptoms of adult forms of DM1 are under development, but their potential role at the level of the nervous system and in particular in forms of CDM1 (which appears to be a distinct disorder of neuronal development) is also to be clarified.

To this end, a better definition of neurocognitive profiles and their evolution is essential for the purposes of evaluating the effectiveness of experimental therapies.

DETAILED DESCRIPTION:
A. Recruitment of patients with a defined diagnosis of Myotonic Dystrophy type 1 (see following inclusion and exclusion criteria)

B) Clinical and cognitive evaluation

1. neurological and neuromuscular examination, compilation of the MIRS-muscle scale and EPWORTH scale-daytime sleepiness (1 session of approximately 1 hour);
2. administration of a neuropsychological battery, in order to define the level of cognitive functioning and to frame a detailed function-specific profile (multiple sessions to be defined based on the collaboration of the patients) investigating the following areas:

   1. intelligence quotient;
   2. attention;
   3. memory;
   4. visual-constructive skills and executive functions
3. psychiatric examination and administration of psychological tests (MMPI-2, Minnesota Multiphasic Personality Inventory 2) to investigate any psychopathologies (behavioral disorders, anxiety disorders, developmental disorders, hyperactivity/attention deficit) and to define the psychological-behavioral profile and adaptive (Vineland Adaptive Behavioral Scale)
4. neuroimaging examination through Morphological magnetic resonance and Diffusor Tensor imaging and Voxel Based Morphometry protocols
5. based on the clinical conditions, a cardiological evaluation will also be carried out (including instrumental tests such as Electrocardiogram ECG, echocardiogram and 24-hour ECG) and pneumological evaluation (with recording of nocturnal oximetry, spirometry), eye examination, phoniatric examination and logopedic evaluation (aimed at evaluating chewing/swallowing)

ELIGIBILITY:
Inclusion criteria:

1. genetically defined diagnosis of Steinert myotonic dystrophy
2. age <35 years
3. reading and signing the informed consent. For the congenital form: presence of hypotonia and weakness at birth, for the juvenile form: onset between 1 and 10 years with normal pre-perinatal history.

Exclusion criteria

1. other concomitant pathologies that completely prevent the execution of clinical assessments
2. presence of devices and prostheses that prevent the execution of the MRI
3. lack of family compliance. -

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a defined diagnosis of MYotonic Dystrophy type 1, congenital and juvenile form
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Motor function evaluation by Muscular Impairment Rating Scale | through study completion,an average of 2 years
  Muscular Impairment Rating Scale (MIRS) in assessing patients with myotonic dystrophy type 1 (DM1). The MIRS is a ordinal five-point rating scale, where grade 1 = no clinical muscular impairment; grade 2 = early muscular impairment (clinical myotonia, facial weakness, and weakness of neck flexors) without limb weakness; grade 3 = distal weakness; grade 4 = mild to moderate (3 ≤ core < 5) proximal weakness; grade 5 = severe (MRC score<3)proximal weakness proximal weakness
cognitive evaluation by Wechsler Intelligence scale | through study completion,an average of 2 years
  Wechsler Intelligence scale: mean score 100 SD 15 (SD: Standard Deviation):deficiency when 2 Standard Deviation below average)
cognitive evaluation by Raven Matrices | through study completion,an average of 2 years
  Raven Matrices , Z scores=/> 0,00 (in range); Z scores =/< -2,00 (deficiency)
cognitive evaluation by Continous Performance Test 3 | through study completion,an average of 2 years
  Continous Performance Test 3: T mean Scores 50 SD 10 (SD: standard deviation) (T=45-59 in range; T =/>60 below range)
cognitive evaluation by Trail Making Test A-B | through study completion,an average of 2 years
  Trail Making Test A-B: Z scores=/> 0,00 (in range); Z scores =/< -2,00 (deficiency)
cognitive evaluation by Digit Span and CORSI Test | through study completion,an average of 2 years
  Digit Span and CORSI Test:Z scores=/> 0,00 (in range); Z scores =/< -2,00 (deficiency)
cognitive evaluation by Rey Figure test | through study completion,an average of 2 years
  Rey Figure test: Z scores=/> 0,00 (in range); Z scores =/< -2,00 (deficiency):

SECONDARY OUTCOMES:
clinical evaluation by Epworth Sleepiness Scale | through study completion,an average of 2 years
  Epworth Sleepiness Scale: scores from 0 to 24; above 10, clinical risk.
cognitive evaluation by Wisconsin Card Sorting Test | through study completion,an average of 2 years
  Wisconsin Card Sorting Test: mean score 100 SD 15 (SD: standard deviation) : deficiency when 2 Standard Deviation below average
cognitive evaluation by Tower of London test | through study completion,an average of 2 years
  Tower of London:mean score 100 SD 15 deficiency when 2 Standard Deviation below average)
cognitive and behavioral evaluation by Minnesota Multiphasic Personality Inventory | through study completion,an average of 2 years
  Minnesota Multiphasic Personality Inventory- MMPI 2: mean score 50 SD 10 ((SD: standard deviation)
cognitive and behavioral evaluation by Vineland Adaptive Behavior Scales | through study completion :an average of 2 years
  Vineland Adaptive Behavior Scales mean score 100 SD 15 (SD: standard deviation) :deficiency when 2 Standard Deviation below average

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Grazia D'Angelo, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No